CLINICAL TRIAL: NCT00481377
Title: Ablation for ICD Intervention Reduction in Patients With CAD - a Prospective Randomized Trial
Brief Title: Ablation for ICD Intervention Reduction in Patients With CAD
Acronym: ABLATION 4 ICD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IK-NP-0021-42/1013/07
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2008-07-21 (Estimated); Status verified 2008-07

CONDITIONS: Ventricular Tachycardia; Coronary Artery Disease; Implantable Cardioverter-Defibrillator
Keywords: Ablation; Ventricular tachycardia; coronary artery disease; Implantable cardioverter defibrillator interventions
MeSH Terms: conditions — Tachycardia, Ventricular; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ablation

SUMMARY:
The aim of this study is to assess the role of ablation in appropriate ICD interventions reduction in patients with coronary artery disease. The group will consist of 200 patients with implanted ICD and appropriate intervention in the 3 months prior to enrollment. The patients will be randomized into ablation arm and conventional treatment. Number of appropriate ICD interventions is the primary endpoint of this study. All patients will have control follow-up visits every 3 months. The follow-up will be based on ICD memory.

ELIGIBILITY:
Inclusion Criteria:

* Coronary Artery Disease
* ICD implanted
* Appropriate ICD intervention during the 3 months prior to enrollment
* Coronary angiography during the 6 months prior to enrollment
* Possible revascularization
* Age over 18 years
* Signed informed consent

Exclusion Criteria:

* Age less then 18 years
* Pregnancy
* Active participation in other trial
* Heart failure (NYHA IV)
* Contraindications for ablation procedure: i.e. left ventricular thrombus, artificial aortic or mitral valve, no vascular access.
* Monomorphic, incessant, ventricular tachycardia
* Revascularization or other cardio-surgical procedure scheduled in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-05; Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Number of appropriate ICD interventions

SECONDARY OUTCOMES:
Overall mortality
Cardiac mortality
Hospitalization due to arrhythmia or heart failure
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz J Szumowski, MD, PhD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, Warsaw, Masovian Voivodeship, Poland

REFERENCES:
- [Derived] Szumowski L, Przybylski A, Maciag A, Derejko P, Bodalski R, Zakrzewska J, Orczykowski M, Szufladowicz E, Szwed H, Walczak F. Outcomes of a single centre registry of patients with ischaemic heart disease, qualified for an RF ablation of ventricular arrhythmia after ICD intervention. Kardiol Pol. 2009 Feb;67(2):123-7; discussion 128-9. English, Polish. PMID 19288374